CLINICAL TRIAL: NCT03528369
Title: A Phase 2 Double-Blind Clinical Trial to Examine the Comparative Effects on Osteoarthritic Knee Pain of CGS-200-1 (1% Capsaicin Topical Liquid), CGS-200-5 (5% Capsaicin Topical Liquid), and CGS-200-0 (Vehicle, No Capsaicin)
Brief Title: A Phase 2 Clinical Trial Examining the Effects on Osteoarthritic Knee Pain of CGS-200-1, CGS-200-5 and Vehicle Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Propella Therapeutics (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VZU00025
Record Dates: First submitted 2018-03-20; First posted 2018-05-17 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CGS-200-1 (Experimental): CGS-200-1 (1% Capsaicin content), a topical analgesic liquid. A single dose will be topically applied to both knees for 60 minutes on Visit 2 on Day 1, Day 2, Day 3, and Day 4.
  Interventions: Drug: CGS-200-1
- CGS-200-5 (Experimental): CGS-200-5 (5% Capsaicin content), a topical analgesic liquid. A single dose will be topically applied to both knees for 60 minutes on Visit 2 on Day 1, Day 2, Day 3, and Day 4.
  Interventions: Drug: CGS-200-5
- CGS-200 Vehicle (Sham Comparator): CGS-200 Vehicle (no Capsaicin), a topical liquid. A single dose will be topically applied to both knees for 60 minutes on Visit 2 on Day 1, Day 2, Day 3, and Day 4.
  Interventions: Drug: CGS-200 Vehicle

INTERVENTIONS:
Drug: CGS-200-1 — CGS-200-1 is a multi-component formulation in which the active ingredient for the intended therapeutic effect is capsaicin at a level of 1% for this study.
  Other Names: CGS-200 (1% capsaicin)
  Arms: CGS-200-1
Drug: CGS-200-5 — CGS-200-5 is a multi-component formulation in which the active ingredient for the intended therapeutic effect is capsaicin at a level of 5% for this study.
  Other Names: CGS-200 (5% capsaicin)
  Arms: CGS-200-5
Drug: CGS-200 Vehicle — CGS-200 Vehicle contains all of the ingredients in CGS-200-1 and CGS-200-5 except for capsaicin.
  Other Names: CGS-200 (0% capsaicin)
  Arms: CGS-200 Vehicle

SUMMARY:
This is a multi-center, randomized, double-blind clinical trial to examine the comparative effects on OAKP of CGS-200-1 (1% Capsaicin content) (N=40), CGS-200-5 (5% Capsaicin content) (N=40), and CGS-200 Vehicle (no Capsaicin) (N=40) in subjects with OA of the knees according to the 1986 American College of Rheumatology (ACR) criteria. Assigned doses will be applied at the clinic for 60 minutes on each of four consecutive days.

DETAILED DESCRIPTION:
Subjects will be randomized to one of the three Arms in this study: CGS-200-1 or CGS-200-5 or CGS-200 Vehicle (CGS-200-0). All subjects will receive 4 consecutive days of treatment and will then be followed up until the Day 94 visit.

Even though both knee(s) will receive application of study test materials, with regard to reduction in WOMAC pain and VAS pain score associated with study treatments, only one knee will be indicated as the "Study Knee". This will be the knee with the highest WOMAC pain score at screening. If both knees have equal WOMAC pain scores at baseline, then the right knee will be considered the "Study Knee" with regard to WOMAC pain and VAS pain score reduction.

Data will be collected from Day 1 through Day 5 and then again on Days 19, 35, 64 and 94 for efficacy, tolerability, and safety measures. The Investigators, all site staff and Clinical Research Organization (CRO) personnel (except the Medical Monitor providing safety oversight) directly involved in the study will remain blinded to the treatment assignment throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis (OA) of both knees;
* OA of both knees must be confirmed by tibiofemoral joint radiographs obtained within the past 6 months;
* Rheumatoid factor (RF) negative and Erythrocyte sedimentation rate (ESR) <40 mm/hr;
* Chronic knee pain in at least 1 knee for > 3 months;
* WOMAC pain score of > 250 (using VAS WOMAC format) at screening, and at baseline, in at least one knee;
* Knee pain score of > 5 on the NRS pain scale at screening, and at baseline, in at least one knee;
* Knee pain is not potentially due to acute trauma unrelated to OA (no acute traumatic knee injury in medical history);
* No burning-stinging pain, unrelated to subject's knee pain, at intended site of application;
* Knee pain must be greater than pain in any other part of subject's body;
* American College of Rheumatology (ACR) global functional status I, II, or III (excluding IV).

Exclusion Criteria:

* Spontaneously improving or rapidly deteriorating OA of the knee;
* Rheumatoid or psoriatic arthritis, or a form of arthritis (e.g. gout, pseudogout), Paget's disease of bone, or any other disease affecting the joints that are inconsistent with a diagnosis of idiopathic OA;
* Labile or poorly controlled hypertension;
* Use of steroids for 1 month prior to screening, or intraarticular-visco-supplementation within 3 months prior to screening;
* Used any capsaicin-containing product on or in the vicinity of the knee within 4 weeks prior to screening;
* Used topically applied products (including emollients or moisturizers) on or in the vicinity of the knees or shaved the knees within 2 days prior to the first application of study drug; or an open wound near the knee; cutaneous erythema or edema; any inflammatory skin lesions such as eczema or psoriasis; cutaneous infections; or any other compromise of the skin;
* Requires or anticipates any surgical procedure within 3 months prior to screening, has had surgery on the affected joint within 6 months prior to screening, has a prosthesis in either knee, or would require surgery while participating in the trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Clinical Operations, Study Director — Vizuri Health Sciences
Locations (6):
- United States (6):
  - Clinical Research of West Florida, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - McIlwain Medical Group, Tampa, Florida
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Radiant Research, Inc., Dallas, Texas
  - Radiant Research, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 6 investigative sites in the US.
Pre-assignment Details: Subjects were randomized to receive one of three treatments after the investigator deemed them to qualify for the study.
Period: Overall Study
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Started | 40 | 42 | 40
Completed | 37 | 41 | 40
Not Completed | 3 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle | Total
Number analyzed (Participants) | 40 | 42 | 40 | 122
Age, Continuous [Mean (Full Range); unit: years] | 59.4 [41 to 75] | 61.1 [44 to 74] | 59.5 [40 to 72] | 60 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 24 | 77
  Male | 11 | 18 | 16 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 10 | 8 | 20
  Not Hispanic or Latino | 38 | 32 | 32 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 9 | 17 | 37
  White | 28 | 33 | 22 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 42 | 40 | 122
Baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score [Mean (Full Range); unit: units on a scale] — The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score is 5 questions relating to pain that the subject responds to using a 100mm visual analogue scale. The minimum score is 0 and the maximum score is 500. The higher the number the worse the outcome.
  units on a scale | 357.0 [260 to 486] | 350.7 [266 to 460] | 346.8 [254 to 490] | 351.5 [254 to 490]

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score From Baseline to Day 35
Description: The Primary Efficacy endpoint of this study will be to examine the extent of change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score, relative to baseline, provided by once daily, one-hour application of Vehicle (CGS-200-0), CGS-200-1 and CGS-200-5 at Baseline (< 30 minutes prior to first daily application) and Day 35 (31 days after fourth daily application).
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score is 5 questions relating to pain that the subject responds to using a 100mm visual analogue scale. The minimum score is 0 and the maximum score is 500. Reduction in pain is expressed as a difference from baseline to Study Day 35. Positive numbers indicate increases and negative numbers indicate decreases. .
Time Frame: 35 days after the last dose of study drug on Day 4
Population: All subjects that received at least one dose of study drug and had at least one evaluable post-dosing efficacy endpoint.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 39 | 40 | 39
units on a scale | -130.7 [-354 to 54] | -159.7 [-376 to 34] | -99.0 [-328 to 73]

2. Secondary Outcome: Secondary Efficacy Endpoint #1: Extent of Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score From Baseline to Day 5, 19, 64 and 94.
Description: The extent of change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score, relative to baseline, provided by once daily, one-hour application of CGS-200-0, CGS-200-1 and CGS-200-5 from Baseline to Day 5, 19, 64 and Day 94.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score is 5 questions relating to pain that the subject responds to using a 100mm visual analogue scale. The minimum score is 0 and the maximum score is 500. Positive numbers indicate increases and negative numbers indicate decreases.
Time Frame: Days 5, 19, 65 and 94 after the last dose of study drug on Day 4
Population: All subjects who received at least one dose of study drug. Differences in subjects is due to subjects who withdrew from the study prior to the efficacy assessment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 40 | 42 | 40
units on a scale
  Day 5 WOMAC Pain Score Change from Baseline: number analyzed (Participants) | 40 | 41 | 40
  Day 5 WOMAC Pain Score Change from Baseline | -113.1 [-359 to 42] | -157.5 [-367 to 40] | -64.5 [-409 to 57]
  Day 19 WOMAC Pain Score Change from Baseline | -131.8 [-338 to 75] | -171.7 [-388 to 21] | -66.4 [-289 to 72]
  Day 64 WOMAC Pain Score Change from Baseline | -79.5 [-345 to 132] | -169.8 [-358 to 34] | 75.4 [-291 to 107]
  Day 94 WOMAC Pain Score Change from Baseline: number analyzed (Participants) | 37 | 39 | 40
  Day 94 WOMAC Pain Score Change from Baseline | -111.8 [-349 to 72] | -147.6 [-378 to 98] | -80.1 [-332 to 90]

3. Secondary Outcome: Patient Reported Burning-Stinging Pain (BSP) During Application of Study Drug.
Description: The average amount of burning-sting pain as reported by the subject using a 0 - 10 numerical rating scale (NRS). Higher scores indicate more pain.
Time Frame: 60 minutes after study drug application on Study Days 1,2,3,4
Population: All subjects who have received at least one dose of study drug. The number of subjects analyzed differs in some cases due to missing data.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 40 | 42 | 40
units on a scale
  Mean Burning-Stinging Pain on Day 1 | 1.36 [0 to 7.75] | 2.70 [0 to 7.25] | 0.36 [0 to 3.25]
  Mean Burning-Stinging Pain on Day 2: number analyzed (Participants) | 40 | 40 | 39
  Mean Burning-Stinging Pain on Day 2 | 0.75 [0 to 3.75] | 1.71 [0 to 7.75] | 0.49 [0 to 5.75]
  Mean Burning-Stinging Pain Day 3: number analyzed (Participants) | 40 | 40 | 39
  Mean Burning-Stinging Pain Day 3 | 0.70 [0 to 3.50] | 1.53 [0 to 7.25] | 0.22 [0 to 2.50]
  Mean Burning-Stinging Pain Day 4 | 0.56 [0 to 2.50] | 1.47 [0 to 7.00] | 0.20 [0 to 3.00]

4. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index Stiffness Scores.
Description: Day 5, 19, 35, 64 and 94 Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index Stiffness Scores.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score is 2 questions relating to stiffness that the subject responds to using a 100mm visual analogue scale. The minimum score is 0 and the maximum score is 200. Positive numbers indicate increases and negative numbers indicate decreases.
Time Frame: Day 5, 19, 35, 64 and 94 days after the last dose of study drug on Study Day 4
Population: All subjects that received at least one dose of study drug and had at least one evaluable post-dosing efficacy endpoint. Differences in number of subjects is due to subjects early withdrawal from the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 40 | 42 | 40
units on a scale
  Day 5 WOMAC Stiffness Score Change from Baseline: number analyzed (Participants) | 40 | 41 | 40
  Day 5 WOMAC Stiffness Score Change from Baseline | -50.7 [-147 to 58] | -59.6 [-166 to 32] | -25.6 [-188 to 39]
  Day 19 WOMAC Stiffness Score Change from Baseline: number analyzed (Participants) | 39 | 40 | 39
  Day 19 WOMAC Stiffness Score Change from Baseline | -52.2 [-152 to 109] | -65.5 [-161 to 65] | -26.8 [-152 to 29]
  Day 35 WOMAC Stiffness Score Change from Baseline: number analyzed (Participants) | 39 | 40 | 39
  Day 35 WOMAC Stiffness Score Change from Baseline | -46.0 [-154 to 78] | -54.8 [-137 to 33] | -39.8 [-158 to 30]
  Day 64 WOMAC Stiffness Score Change from Baseline: number analyzed (Participants) | 38 | 40 | 39
  Day 64 WOMAC Stiffness Score Change from Baseline | -32.2 [-150 to 114] | -59.5 [-162 to 29] | -28.1 [-158 to 42]
  Day 94 WOMAC Stiffness Score Change from Baseline: number analyzed (Participants) | 37 | 39 | 40
  Day 94 WOMAC Stiffness Score Change from Baseline | -42.7 [-151 to 37] | -56.8 [-166 to 45] | -31.9 [-159 to 42]

5. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index Function Scores.
Description: Day 5, 19, 35, 64 and 94 Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index Function Scores.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function score is 17 questions relating to physical function that the subject responds to using a 100mm visual analogue scale. The minimum score is 0 and the maximum score is 1700. Positive numbers indicate increases and negative numbers indicate decreases.
Time Frame: Day 5, 19, 35, 64 and 94 days after the last dose of study drug on Study Day 4
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 40 | 42 | 40
units on a scale
  Day 5 WOMAC Function Score Change from Baseline: number analyzed (Participants) | 40 | 41 | 40
  Day 5 WOMAC Function Score Change from Baseline | -385.0 [-1174 to 346] | -499.0 [-1397 to 59] | -198.1 [-1343 to 223]
  Day 19 WOMAC Function Score Change from Baseline: number analyzed (Participants) | 39 | 40 | 39
  Day 19 WOMAC Function Score Change from Baseline | -398.7 [-1275 to 501] | -583.7 [-1415 to 100] | -192.1 [-1219 to 315]
  Day 35 WOMAC Function Score Change from Baseline: number analyzed (Participants) | 39 | 40 | 39
  Day 35 WOMAC Function Score Change from Baseline | -367.8 [-1240 to 456] | -523.0 [-1397 to 286] | -296.9 [-1278 to 279]
  Day 64 WOMAC Function Score Change from Baseline: number analyzed (Participants) | 38 | 40 | 39
  Day 64 WOMAC Function Score Change from Baseline | -218.9 [-1286 to 796] | -515.9 [-1261 to 299] | -213.7 [-901 to 357]
  Day 94 WOMAC Function Score Change from Baseline: number analyzed (Participants) | 37 | 39 | 39
  Day 94 WOMAC Function Score Change from Baseline | -337.5 [-1273 to 249] | -506.5 [-1406 to 191] | -233 [-1297 to 349]

6. Other Pre Specified Outcome: Number of Subjects With Skin Reactions of Erythema or Pruritus.
Description: Investigator reports of erythema or pruritus at the site of study drug application.
Time Frame: Study Day 1 through Study Day 35 after the first application of study drug (Study Day 1)
Population: All subjects who have received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 40 | 42 | 40
participants
  Erythema | 1 | 1 | 0
  Pruritus | 2 | 2 | 0

7. Other Pre Specified Outcome: Number of Subjects With Durability of Efficacy Response
Description: Subjects who had a clinical response (i.e., reduction of at least 50% in WOMAC pain score) at the Day 5 visit and who remained at this reduction of pain score or lower at Days 19, 35, 64, and the Day 94 visit were considered to have a durable clinical response through Day 94. Subjects who had a clinical response at no more than one of the post Day 5 visits were considered to have a durable response through the last day at which reduction in WOMAC pain score is at least 50%. Subjects who had less than 50% WOMAC pain score reduction on two or more of the post Day 5 visits were considered to have failed to achieve a durable clinical response.
Time Frame: Days 35, 64 and 94 day after the last dose of study drug on Study Day 4
Population: All subjects that received at least one dose of study drug and had at least one evaluable post-dosing efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 40 | 42 | 40
Participants
  Day 35: number analyzed (Participants) | 40 | 41 | 40
  Day 35: Responders | 15 | 19 | 11
  Day 35: Non-Responders | 25 | 22 | 29
  Day 64 Responders: number analyzed (Participants) | 40 | 41 | 40
  Day 64 Responders: Responders | 5 | 23 | 9
  Day 64 Responders: Non-Responders | 35 | 18 | 31
  Day 94 Responders: number analyzed (Participants) | 40 | 41 | 40
  Day 94 Responders: Responders | 10 | 18 | 10
  Day 94 Responders: Non-Responders | 30 | 23 | 30

8. Post Hoc Outcome: Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index Total Scores (Pain, Stiffness and Function).
Description: Day 5, 19, 35, 64 and 94 Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index total scores (pain, stiffness and function) from Baseline.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score is 24 questions relating to pain, stiffness and physical function that the subject responds to using a 100mm visual analogue scale. The minimum score is 0 and the maximum score is 2400. Positive numbers indicate increases and negative numbers indicate decreases.
Time Frame: Day 5, 19, 35, 64 and 94 days after the last dose of study drug on Study Day 4
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
Number analyzed (Participants) | 40 | 42 | 40
units on a scale
  Day 5 WOMAC Total Score Change from Baseline: number analyzed (Participants) | 40 | 41 | 40
  Day 5 WOMAC Total Score Change from Baseline | -548.8 [-1747 to 572] | -716.1 [-1928 to 22] | -288.1 [-1940 to 285]
  Day 19 WOMAC Total Score Change from Baseline: number analyzed (Participants) | 39 | 40 | 39
  Day 19 WOMAC Total Score Change from Baseline | -582.8 [-1747 to 572] | -820.9 [-1961 to 121] | -285.3 [-1660 to 406]
  Day 35 WOMAC Total Score Change from Baseline: number analyzed (Participants) | 39 | 40 | 39
  Day 35 WOMAC Total Score Change from Baseline | -544.5 [-1748 to 366] | -737.5 [-1899 to 353] | -435.8 [-1747 to 370]
  Day 64 WOMAC Total Score Change from Baseline: number analyzed (Participants) | 38 | 40 | 39
  Day 64 WOMAC Total Score Change from Baseline | -330.6 [-1781 to 901] | -745.2 [-1759 to 337] | -317.2 [-1261 to 506]
  Day 94 WOMAC Total Score Change from Baseline: number analyzed (Participants) | 37 | 39 | 39
  Day 94 WOMAC Total Score Change from Baseline | -491.9 [-1769 to 331] | -710.8 [-1939 to 314] | -345.9 [-1769 to 331]

ADVERSE EVENTS:
Time Frame: AEs were captured from start of study drug treatment through Day 94
Description: Severity was graded using the Rheumatology Common Toxicity Criteria (RCTC) version 2.0
Arm/Group | CGS-200-1 | CGS-200-5 | CGS-200 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 36/40 | 41/42 | 24/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGS-200-1 (N=40) | CGS-200-5 (N=42) | CGS-200 Vehicle (N=40)
Application Site Pain (General disorders) | 30 (30) | 40 (40) | 20 (20)
Application site paraesthesia (General disorders) | 2 (2) | 4 (4) | 2 (2)
Application site pruritus (General disorders) | 3 (3) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results and communications prior to public release, and Sponsor can embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to the Sponsor for review. At all times, PIs retain editorial control of all publications and have a right to publish the study data, subject only to Sponsor's time-limited right to protect its intellectual property rights and prevent disclosure of Sponsor's confidential information.

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03528369/Prot_001.pdf
  • Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT03528369/SAP_000.pdf